CLINICAL TRIAL: NCT00728182
Title: A Phase II, Multicenter, Randomized, Fasting, Double-Blind, Placebo-Controlled, Safety, Tolerability and Efficacy Study Evaluating a Single Dose of Intravenous NA-1 in Male and Female Patients Undergoing Endovascular Repair of Brain Aneurysms
Brief Title: Evaluating Neuroprotection in Aneurysm Coiling Therapy
Acronym: ENACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Collaborators: Arbor Vita Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3302 (NA-1-002)
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-08

CONDITIONS: Stroke
Keywords: Stroke; Vascular cognitive impairment; Coiling; Endovascular repair; Brain aneurysm; NA-1
MeSH Terms: conditions — Stroke; Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NA-1 (Experimental): 20 amino acid peptide that consists of a 9 amino acid domain that inhibits PSD-95 and a 11 amino acid domain than enables the peptide to cross the blood-brain barrier.
  Interventions: Drug: NA-1
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NA-1 — single intravenous dose of 2.6 mg/kg of NA-1 administered as a 10-minute infusion
  Arms: NA-1
Drug: Placebo — single intravenous dose of 2.6 mg/kg of placebo administered as a 10-minute infusion
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose, design investigating the safety, tolerability and efficacy of NA-1, a peptide designed to reduce ischemic brain damage. Up to 200 male and female patients undergoing endovascular repair of brain aneurysm will be dosed with 2.60 mg/kg of NA-1 or placebo as a 10 minute intravenous infusion after completion of the endovascular procedure on Day 1 of the study period. Subjects will undergo interim procedures Days 2-4 and end-of study procedures on Day 30. Standard safety criteria will be analysed. Efficacy endpoints include the ability of NA-1 to: 1) reduce the volume of ischemic embolic strokes, 2) reduce the number of ischemic embolic strokes, 3) reduce vascular cognitive impairment, and 4) reduce the frequency of large strokes induced by the endovascular procedure. The plasma concentrations of NA-1 will also be analyzed.

ELIGIBILITY:
Inclusion Criteria

* A diagnosis of a ruptured or unruptured brain aneurysm deemed suitable for repair by neuroendovascular techniques involving intraluminal occlusion by detachable platinum coils, stent-assisted coiling, pipeline stent, balloon-assisted coiling, covered stent only, neck-bridge device, re-coiling, or re-treatment of a previously coiled/treated aneurysm. There are no restrictions on adjunctive devices. For patients with a ruptured aneurysm, endovascular repair must take place within 72 hours of the ictal haemorrhage.
* If the aneurysm has ruptured, patient should be Grade I-III on the World Federation of Neurological Surgeons (WFNS) grading scale for subarachnoid hemorrhage. If the patient is intubated but alert and able to follow commands (at least a 2-step command), and is not kept intubated for neurological status (i.e., WFNS Grade IV or V), the patient is considered WFNS Grade III and is eligible for the trial.
* Absence of ongoing ischemic symptoms such as transient ischemic attacks, minor strokes, stroke-in-evolution, or clinical evidence of cerebral vasospasm within 2 weeks prior to randomization. (If a CT scan, cerebral angiogram, or other imaging performed during the 2 weeks prior to randomization shows radiological vasospasm deemed by the treating physician to be potentially clinically significant, the subject is excluded.)
* Brain MRI imaging (DWI and FLAIR sequences) within 2 weeks prior to the endovascular aneurysm repair procedure as detailed in Section 8.2. Imaging must not demonstrate any focal ischemic stroke defined as a new region of restricted diffusion and/or a focal area of reduced perfusion on a relative mean transit time (rMTT) or relative time to peak (rTTP) map
* Male or female with a minimum age of 18 years on the day of enrolment.
* Female subjects of childbearing potential: Negative pregnancy test. After enrolment, blood will be drawn from women of childbearing potential for a confirmatory test of pregnancy as evaluated by a serum B-hCG test. The definition of non-childbearing potential includes the following:

  * Surgically sterile (e.g., hysterectomy with or without oophorectomy; fallopian tube ligation; endometrial ablation), at least 30 days prior to signature of the Informed Consent form
  * At least 5 years post-menopause (i.e., 6 years post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing. Non-surgically sterile females or females with undocumented post-menopausal status must be willing to use a medically approved method of birth control for 3 months after completion of dosing.
* Non-surgically sterile males or males with partners of childbearing potential must be willing to use condoms with spermicide for 3 months after completion of dosing.
* Body weight less than or equal to 180 kg.
* Normal or abnormal but not clinically significant findings in the

  * non-neurological physical examination
  * 12-lead ECG
  * PQ or PR interval less than or equal to 210 msec;
  * In unruptured aneurysm cases, QTc interval less than 450 msec for males or 470 msec for females. For ruptured aneurysm cases, QTc interval is not restricted.
  * vital signs
  * blood pressure between 80-180/50-100 mm Hg,
  * body temperature less than or equal to 38.5oC
* Informed consent and availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.

Exclusion Criteria

* Dissecting or mycotic brain aneurysm. Fusiform or atherosclerotic intracerebral aneurysms may be eligible for the trial if endovascular treatment is planned with a goal of exclusion of the aneurysm from the circulation.
* Planned endovascular vessel sacrifice as the primary modality for aneurysm treatment.
* Known history of life-threatening allergic reaction to any medication.
* Chronic renal disease defined as a baseline serum creatinine > 150 umol/L.
* Women who are pregnant, or have a positive urine or blood (β-hCG) pregnancy test.
* Women who are breastfeeding.
* Any clinically significant psychiatric or psychological disease, which would preclude the patient from completing the protocol.
* Pre-morbid (estimated) modified Rankin scale score of greater than 2.
* Previous serious traumatic brain injury that would preclude the patient from completing the protocol or preclude MRI analysis of small strokes.
* Patients with known HIV infection.
* Patients who are unable to have an MRI scan for any reason.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study. Previous participation in the ENACT trial (e.g,, to treat a prior aneurysm), participation in another trial involving NA-1 or prior receipt of NA-1.
* Any other medical condition that the site investigator deems would put the patient at excessive risk of participation in the study or an expected life expectancy less than 1 year or that would result in inability to collect clinical outcomes at 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hill, M.D., Principal Investigator — Foothills Medical Centre, University of Calgary
Locations (14):
- United States (3):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Stanford University Medical Center, Stanford, California
  - Oregon Health and Science University, Portland, Oregon
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - QEII Health Sciences Centre - Halifax Infirmary, Halifax, Nova Scotia
  - Hamilton Health Sciences General Site, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hôpital Notre-Dame du Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hopital de l'Enfant Jesus, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Hill MD, Martin RH, Mikulis D, Wong JH, Silver FL, Terbrugge KG, Milot G, Clark WM, Macdonald RL, Kelly ME, Boulton M, Fleetwood I, McDougall C, Gunnarsson T, Chow M, Lum C, Dodd R, Poublanc J, Krings T, Demchuk AM, Goyal M, Anderson R, Bishop J, Garman D, Tymianski M; ENACT trial investigators. Safety and efficacy of NA-1 in patients with iatrogenic stroke after endovascular aneurysm repair (ENACT): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2012 Nov;11(11):942-50. doi: 10.1016/S1474-4422(12)70225-9. Epub 2012 Oct 8. PMID 23051991
- [Derived] Ganesh A, Goyal M, Wilson AT, Ospel JM, Demchuk AM, Mikulis D, Poublanc J, Krings T, Anderson R, Tymianski M, Hill MD; ENACT Trial Investigators. Association of Iatrogenic Infarcts With Clinical and Cognitive Outcomes in the Evaluating Neuroprotection in Aneurysm Coiling Therapy Trial. Neurology. 2022 Apr 5;98(14):e1446-e1458. doi: 10.1212/WNL.0000000000200111. Epub 2022 Feb 15. PMID 35169007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 16, 2008 and March 30, 2011, subjects were recruited to 10 hospitals in Canada and 3 in the United States.
Pre-assignment Details: 12 subjects were randomized into study but did not receive drug:5 due to do endovascular aneurysm repair, 3 due to inability to obtain a pre-procedure MRI,2 due to pre-procedure ECG showing a QTc interval > 450 ms, 1 due to a fatal aneurysm rupture before drug, and 1 due to refusal by anesthesiologist to give drug to a subject with severe COPD.
Groups:
- 1 NA-1: 20 amino acid peptide that consists of a 9 amino acid domain that inhibits PSD-95 and a 11 amino acid domain than enables the peptide to cross the blood-brain barrier.
  NA-1 : single intravenous dose of 2.6 mg/kg of NA-1 administered as a 10-minute infusion
- 2 Placebo: Placebo : single intravenous dose of 2.6 mg/kg of placebo administered as a 10-minute infusion
Period: Overall Study
Arm/Group | 1 NA-1 | 2 Placebo
Started | 92 | 93
Completed | 89 | 90
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 0 | 2
Not completed — Protocol Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 NA-1 | 2 Placebo | Total
Number analyzed (Participants) | 92 | 93 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 78 | 148
  >=65 years | 22 | 15 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 57.72 (10.6) | 56.05 (10.3) | 56.88 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 132
  Male | 28 | 25 | 53
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27
  Canada | 80 | 78 | 158

OUTCOME MEASURES:

1. Primary Outcome: Volume of New FLAIR Lesions(MRI)
Description: Volume of new ischemic lesions as defined by FLAIR MRI at 12-95 hours postdose
Time Frame: Enrolment, Days 2-4
Population: All study patients who received study drug and an analyzable MRI at 12-95 hours postdose.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 91 | 93
mm^3 | 915 (5598) | 477 (1611)
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Comparison of the summed volume of new FLAIR lesions in the NA-1 and placebo treated groups; Test type: Superiority or Other; p = 0.445, ANCOVA; Data were cubic root transformed and modelled with multiple linear regression

2. Secondary Outcome: Number of New DWI Lesions (MRI)
Description: Number of new ischemic lesions as defined by DWI MRI at 12-95 hours postdose.
Time Frame: Enrolment, Day 2-4
Population: All patients who received study drug and an analyzable MRI at 12-95 hours postdose.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 91 | 93
Lesions | 4.1 (6.8) | 7.3 (12.6)
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Comparison of the total number of new ischemic lesions on DWI for NA-1 versus placebo treated groups; Test type: Superiority or Other; p = 0.018, Generalized linear model; With log link and negative bnomial distribution; Adjusted Incidence Rate Ratio = 0.53, 95% CI 2-sided [0.38 to 0.74]

3. Secondary Outcome: Number of New FLAIR Lesions (MRI)
Description: Number of new ischemic lesions as defined by FLAIR MRI at 12-95 hours postdose.
Time Frame: Enrolment, Days 2-4
Population: All patients who received study drug and an analyzable MRI scan at 12-95 hours postdose.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 91 | 93
Lesions | 3.0 (4.4) | 4.8 (7.7)
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Comparison of the total number of new FLAIR lesions in the NA-1 versus placebo treated groups; Test type: Superiority or Other; p = 0.048, Generalized linear model; With log link and negative binomial distribution; Adjusted Incidence Rate Ratio = 0.59, 95% CI 2-sided [0.42 to 0.83]

4. Secondary Outcome: Volume of New DWI Lesions (MRI)
Description: Volume of new DWI lesions as defined by MRI at 12-95 hours postdose.
Time Frame: Enrolment, Days 2-4
Population: All patients who received study drug and an analyzable MRI at 12-95 hours postdose.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 91 | 93
mm^3 | 966 (5266) | 645 (1382)
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Comparison of the summed volume of new ischemic lesions on DWI; Test type: Superiority or Other; p = 0.306, ANCOVA; Data were cubic root transformed and modelled with multiple linear regresion

5. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS).
Description: The NIHSS is a standardized neurological method to measure disability and recovery after stroke. Scores range from 0 to 42, with higher scores indicating increasing severity. Scores were dichotomized into 0-1 (good outcome) versus 2 or above. The number of participants scoring 0-1 on the NIHSS at Day 30 was compared for both groups.
Time Frame: Enrolment, Day 30
Population: All patients who received study drug and outcome assessment at Day 30.
Measure: Number; unit: No. of participants with NIHSS 0-1
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 92 | 93
No. of participants with NIHSS 0-1 | 86 [0.9 to 1.1] | 83 [0.9 to 1.1]
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Number of patients obtaining a score on the NIHSS of 0-1 at Day 30; Test type: Superiority or Other; p = 0.43, Chi-squared; Relative Risk = 1.0, 95% CI 2-sided [0.9 to 1.1]

6. Secondary Outcome: Modified Rankin Scale (mRS).
Description: The mRS is a measure of global disability that has been widely applied for evaluating recovery from stroke. Scores range from 0 to 6, with higher scores indicating greater disability. A score of 0 indicates no residual symptoms; 1 = no significant disability/able to carry out all usual activities, despite some symptoms; 2 = slight disability; 3 = moderate disability; 4 = moderately severe disability; 5 = severe disability; 6 = death. The number of participants scoring 0-2 on the mRS at Day 30 was compared in both treatment groups.
Time Frame: Enrolment, Day 30
Population: All patients who received study drug and an outcome assessment at Day 30
Measure: Number; unit: No. of participants with mRS 0-2
Arm/Group | 1 NA-1 | 2 Placebo
Number analyzed (Participants) | 92 | 93
No. of participants with mRS 0-2 | 86 [0.9 to 1.1] | 87 [0.9 to 1.1]
Statistical Analysis 1: Comparison: 1 NA-1 vs 2 Placebo; Comparison of the number of patients with mRS scores of 0-2 at Day 30 for NA-1 and placebo treated groups; Test type: Superiority or Other; p = 1.00, Chi-squared; Relative Risk = 1.0, 95% CI 2-sided [0.9 to 1.1]

7. Other Pre Specified Outcome: Volume of New FLAIR Lesions (MRI) - Ruptured Aneurysm Subjects
Description: Volume of new ischemic lesions as defined by FLAIR MRI at 12-95 hours postdose (pre-specified subgroup analysis)
Time Frame: Enrolment, Days 2-4
Population: All subjects who entered the study with a ruptured aneurysm, who received study drug and an analyzable MRI at 12-95 hours postdose.
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- 1 NA-1 - Subjects With Ruptured Aneurysms: 20 amino acid peptide that consists of a 9 amino acid domain that inhibits PSD-95 and a 11 amino acid domain than enables the peptide to cross the blood-brain barrier.
  NA-1 : single intravenous dose of 2.6 mg/kg of NA-1 administered as a 10-minute infusion
- 2 Placebo - Subjects With Ruptured Aneurysms: Placebo : single intravenous dose of 2.6 mg/kg of placebo administered as a 10-minute infusion
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
mm^3 | 205 (495) | 1575 (3229)
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.023, ANCOVA

8. Other Pre Specified Outcome: Number of New DWI Lesions (MRI) - Ruptured Aneuryms Subjects
Description: Number of new ischemic lesions as defined by DWI MRI at 12-95 hours postdose(pre-specified subgroup analysis)
Time Frame: Enrolment, Day 2-4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
Lesions | 3.4 (5.9) | 9.47 (11.6)
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.027, Adjusted Incidence Rate Ratio; Adjusted Incidence Rate Ratio = 0.36, 95% CI 2-sided [0.17 to 0.73]

9. Other Pre Specified Outcome: Number of New FLAIR Lesions (MRI) - Ruptured Aneurysm Subjects
Description: Number of new ischemic lesions as defined by FLAIR MRI at 12-95 hours postdose(pre-specified subgroup analysis)
Time Frame: Enrolment, Day 2-4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
Lesions | 2.4 (4.7) | 6.58 (7.5)
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.046, Generalized linear model; Adjusted Incidence Rate Ratio = 0.36, 95% CI 2-sided [0.17 to 0.75]

10. Other Pre Specified Outcome: Volume of New DWI Lesions (MRI) - Ruptured Aneurysm Subjects
Description: Volume of new DWI lesions as defined by MRI at 12-95 hours postdose(pre-specified subgroup analysis)
Time Frame: Enrolment, Day 2-4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
mm^3 | 277 (528) | 1373 (2267)
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.015, ANCOVA

11. Other Pre Specified Outcome: National Institutes of Health Stroke Scale (NIHSS) - Ruptured Aneurysm Subjects
Description: The NIHSS is a standardized neurological method to measure disability and recovery after stroke. Scores range from 0 to 42, with higher scores indicating increasing severity. Scores were dichotomized into 0-1 (good outcome) versus 2 or above. The number of participants scoring 0-1 on the NIHSS at Day 30 was compared for participants with ruptured aneurysms in both treatment groups(pre-specified subgroup analysis).
Time Frame: Enrolment, Day 30
Population: All subjects who entered the study with a ruptured aneurysm, who received study drug and outcome assessment at Day 30.
Measure: Number; unit: No. of participants with NIHSS 0-1
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
No. of participants with NIHSS 0-1 | 18 | 13
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.02, Chi-squared; Relative Risk = 1.5, 95% CI 2-sided [1.1 to 2.0]

12. Other Pre Specified Outcome: Modified Rankin Scale (mRS)- Ruptured Aneurysm Subjects
Description: The mRS is a measure of global disability that has been widely applied for evaluating recovery from stroke. Scores range from 0 to 6, with higher scores indicating greater disability. A score of 0 indicates no residual symptoms; 1 = no significant disability/able to carry out all usual activities, despite some symptoms; 2 = slight disability; 3 = moderate disability; 4 = moderately severe disability; 5 = severe disability; 6 = death. The number of participants scoring 0-2 on the mRS at Day 30 with ruptured aneurysms was compared in both treatment groups(pre-specified subgroup analysis).
Time Frame: Enrolment, Day 30
Measure: Number; unit: No. of participants with mRS 0-2
Arm/Group | 1 NA-1 - Subjects With Ruptured Aneurysms | 2 Placebo - Subjects With Ruptured Aneurysms
Number analyzed (Participants) | 18 | 19
No. of participants with mRS 0-2 | 17 | 14
Statistical Analysis 1: Comparison: 1 NA-1 - Subjects With Ruptured Aneurysms vs 2 Placebo - Subjects With Ruptured Aneurysms; Test type: Superiority or Other; p = 0.18, Chi-squared; Relative Risk = 1.3, 95% CI 2-sided [0.95 to 1.7]

ADVERSE EVENTS:
Arm/Group | 1 NA-1 | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 9/92 | 14/93
Other Adverse Events (participants affected / at risk) | 83/92 | 85/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 NA-1 (N=92) | 2 Placebo (N=93)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Nervous system (Nervous system disorders) | 3 (3) | 9 (14)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Vascular (Vascular disorders) | 3 (3) | 3 (3)
Administration site (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 NA-1 (N=92) | 2 Placebo (N=93)
Headache (Nervous system disorders) | 42 (47) | 37 (39)
Nausea (Gastrointestinal disorders) | 33 (33) | 27 (28)
Vomiting (Gastrointestinal disorders) | 12 (12) | 8 (8)
Hypotension (Vascular disorders) | 9 (10) | 6 (6)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 10 (10)
Hypertension (Vascular disorders) | 4 (4) | 7 (7)
Eye pain (Eye disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (7)
Fatigue (General disorders) | 1 (1) | 7 (7)
Puncture site pain (General disorders) | 5 (5) | 5 (5)
Urinary tract infection (Infections and infestations) | 7 (7) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Dizziness (Nervous system disorders) | 6 (6) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 5 (5)
Anxiety (Psychiatric disorders) | 3 (3) | 7 (8)
Haematuria (Renal and urinary disorders) | 5 (5) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Haematoma (Vascular disorders) | 6 (6) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall have the right to publish any information after prior submittal to NoNO, where NoNO can request a hold for up to 60 days, provided that no publication shall disclose Proprietary Information other than Data containing the results of the Study. Investigators may not publish in the first 18 months after the close of the trial except within a publication representing all participating clinical sites.